CLINICAL TRIAL: NCT01901510
Title: Panchromoendoscopy Using Oral Indigo Carmine Mixed With Polyethylene Glycol Prep
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, M. Edwyn Harrison, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 12-009897
Record Dates: First submitted 2013-06-03; First posted 2013-07-17 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Colonic Polyps
Keywords: polyp
MeSH Terms: conditions — Colonic Polyps; Polyps | interventions — Indigo Carmine; Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- chromoendoscopy (Active Comparator): The intervention arm will have Indigo carmine added to the colonic preperation to perform chromoendoscopy
  Interventions: Drug: Chromoendoscopy (Indigo Carmine)
- Control (Other): The control arm will have minimal Indigo carmine added to the colonic prep in a concentration which will not be enough to perform chromoendoscopy
  Interventions: Other: Control

INTERVENTIONS:
Drug: Chromoendoscopy (Indigo Carmine) — Indigo Carmine will be added to the colonic prep to attempt indirect chromoendoscopy
  Other Names: Indirect chromoendoscopy; Colonoscopy
  Arms: chromoendoscopy
Other: Control — The control will have minimal Indigo Carmine added to the colonic prep. This will serve to color the solution blue for blinding but not enough to provide significant staining for chromoendoscopy.
  Arms: Control

SUMMARY:
This study first is designed to see what dose of indigo carmine ingested orally mixed with the standard colonoscopy prep is needed to provide adequate staining of the right colon. It then will use this adequate staining concentration of Indigo Carmine to study whether this dye will increase the detection of polyps during colonoscopy.

DETAILED DESCRIPTION:
Colon cancer occurs in 5% of the US population. Currently colon cancer screening is recommended at the age of 50 years old for all patients who are at average risk. Colonoscopy is considered the gold standard test for colon cancer screening. This is partly because colonoscopy not only can detect polyps which are cancer precursors but also can remove them, and thereby detecting cancer and its precursors and preventing cancer. Unfortunately recent data suggest that colonoscopy can miss a significant percentage of polyps, especially on the right side of the colon. It is thought that one of the major reasons for missing polyps in the right side of the colon is the fact that they are flat or sessile serrated adenoma, both of which are more difficult than protruding polyps to identify with ordinary colon preparation and colonoscopes. Chromoendoscopy is the application of dye during colonoscopy to enhance detection of polyps. It has been shown that it improves the detection of polyps and thus has the potential of improving the performance of colonoscopy and increasing the detection of these difficult to detect polyps. It is however cumbersome and time consuming, which has discouraged its use. Indigo carmine, one commonly used dye, is actually FDA approved as a food colorant and can be consumed orally. It is minimally absorbed. In addition it is used intravenously for diagnosis of injuries of the urinary system because it is very rapidly excreted by the kidneys. The investigators believe that taking it orally will be well tolerated, and that any of the dye that is absorbed will be rapidly excreted by the kidneys and thus quickly eliminated without any side effects. Effective staining of the colon with indigo carmine and increased detection of polyps could change the current standard of care for screening for colon cancer.

ELIGIBILITY:
Inclusion criteria:

* Patients presenting for screening or surveillance colonoscopy
* Must be aged 50 to 75 yrs
* Must be able and willing to sign informed consent

Exclusion criteria:

* Known Creatinine >1.2
* Cirrhosis
* Pregnancy or breast feeding
* History of anaphylaxis to any dye
* History of bowel surgery or small bowel obstruction
* History of aspiration
* History of dysphagia
* American Society of Anesthesia class >2
* History of abnormal liver function test in the last year
* History of any degree of cytopenia in the last year

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Dose of indigo carmine needed to provide adequate chromoendoscopy of the right sided colon | 24 hours
  The dose in Indigo Carmine in mg per 1/8 - 1/2 gallon needed to provide adequate staining of the cecum and ascending colon.

SECONDARY OUTCOMES:
Cecal intubation rate | 24 hours
Time to cecal intubation | 24 hours
Withdrawal time | 24 hours
Quality of bowel preparation | 24 hours
  The Boston Bowel Preparation Scale will be used to grade the quality of the colonic prep:
  0 = Unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared.
  1. = Portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen due to staining, residual stool and/or opaque liquid.
  2. = Minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well.
  3. = Entire mucosa of colon segment seen well with no residual staining, small fragments of stool or opaque liquid.
Patient tolerance of indigo carmine solution | 30 days
  The rate side effects experienced in the active arm versus the control arm will be compared to determine if side effects experienced are different in both groups. Known common side effect from the Polyethylene based colonic preparation include:
  Malaise Abdominal distension Anal irritation Nausea Abdominal pain Vomiting Rigors Thirst
Quality of staining of the entire colon | 24 hours
  Chromoendoscopy quality:
  Scoring for 3 areas of the colon will be recorded separately:
  Right sided, transverse, left sided Distribution of staining in each area: 0 none, covering less than 50% = 1, patchy covering more than 50%=2, staining most of the mucosa (>80%) =3
  Intensity of staining: none = 0, poor= 1, fair =visible but not obscuring the vasculature, good= visible and obscuring the vasculature.
Adenoma detection rate | 2 weeks
Total number of non rectal serrated polyps detected | 2 weeks
Total number of sessile serrated adenoma detected | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: M Harrison, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States